CLINICAL TRIAL: NCT03422874
Title: A Phase I Dose Escalation Study of Nelfinavir Plus MLN9708 in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Dose Escalation Study of Nelfinavir Plus MLN9708 in Patients With Advanced Solid Tumors or Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew support
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D14037
Record Dates: First submitted 2015-08-31; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Neoplasms; Lymphoma
Keywords: Advanced Solid Tumors; Lymphoma; Nelfinavir; MLN9708; proteasome inhibitor
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — ixazomib; Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nelfinavir plus MLN9708 (Experimental): Both Nelfinavir and MLN9708 will be given orally (by mouth). MLN9708 will be given as 3 mg orally twice weekly. Study drugs will be administered on 21-day treatment cycles. All cycles are 21 days.
  During the first cycle of MLN9708 only will initially be administered orally at a fixed dose of 3mg twice weekly for 2 weeks, on Mondays and Thursdays during this treatment cycle. During the third week there will be no study combination drug therapy(for Cycle 1 only). During Cycles 2 and 3, MLN9708 administered twice weekly on Mondays and Thursdays for the first 2 weeks of Cycles 2 and 3. Nelfinavir (escalating cohorts [1250mg, 1875mg, 2500mg, 3125mg]) will be administered orally twice daily in the dose cohorts listed.
  Interventions: Drug: MLN9708; Drug: Nelfinavir

INTERVENTIONS:
Drug: MLN9708 — MLN9708 is a second-generation reversible proteasome inhibitor which shows greater oral bioavailability, improved pharmacokinetics and enhanced antitumor activity compared with bortezomib (VELCADE®).
  Other Names: Ixazomib
Drug: Nelfinavir — Nelfinavir is an oral HIV protease inhibitor approved by FDA in 1997, now available in generic form. It has a well established safety profile in HIV patients when administered at the recommended dose of 1250 mg PO BID. Nelfinavir was shown to induce ER stress in cancer cell lines and xenograft tumors leading to apoptosis and tumor growth inhibition.
  Other Names: Viracept

SUMMARY:
This is an open label, dose escalation, phase I study of the combination of MLN9708 plus Nelfinavir.

DETAILED DESCRIPTION:
This is an open label, dose escalation, phase I study of the combination of MLN9708 MLN9708 plus Nelfinavir. It will use a 3+3 cohort design to determine the maximum tolerated dose of the combination, which will be defined as the highest dose cohort where < 1/6 patients develop a dose limiting toxicity. The maximum tolerated dose cohort will be expanded to have at least 6 patients with biopsiable tumors who undergo pretreatment and post treatment tumor biopsies for molecular pharmacodynamic markers.

ELIGIBILITY:
Inclusion Criteria

* Advanced or metastatic, histologically/cytologically confirmed malignant solid tumor or any lymphoma, not expected to clinically benefit from standard therapy.
* Life expectancy greater than 3 months.
* Previous chemotherapy and/or radiotherapy must have been completed at least four weeks before enrollment(six weeks for prior treatment with mitomycin or nitrosoureas) and patients should have recovered from all toxicities of that therapy before treatment under this protocol.
* All patients must have recovered from any surgical procedure.
* Serum creatinine must be within the institutional limits of normal and an estimated creatinine clearance of ≥ 60 mL/min.

Calculated by: Weight (in kg) X (140 - age) / (72 X Serum Creatinine)

* In females, multiply by 0.85. Alternatively, creatinine clearance may be measured from a 24 hour urine collection.
* Total bilirubin <2 x ULN. SGOT/AST and ALT must be less than or equal to 2.5 times the upper limit of institutional normal.
* Hb > 9.0 g/dL and absolute neutrophil count ≥ 1,500/mm3, and platelet count ≥ 100,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
* Patients must be 18 years of age or older.
* Patients must have a Karnofsky Performance Status of >70%
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, sympto-thermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients who:

  * Even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:
  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, sympto-thermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Brain metastases must be treated and stable for at least 3 months before the start of the treatment
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria

* Inability or unwillingness to swallow capsules.
* Patients with active hepatitis B or C.
* Patients with known HIV infection.
* Ongoing or active systemic infection.
* Evidence of current uncontrolled cardiovascular conditions including, but not limited to uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Pregnant or lactating female patients.
* Patients with malabsorption syndromes, or who have undergone a resection or bypass of the distal stomach/ pylorus, or small bowel.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial.
* Use of strong CYP 3A4 or P-gp inhibitors and/or inducers.
* Use of strong CYP 1A2 inhibitors and/or inducers.
* See Table of prohibited drugs (Appendix G).
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* Failure to have fully recovered (i.e., < Grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Major surgery within 14 days before enrollment.
* Radiotherapy within four weeks before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has > Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08-04 (Estimated); Study Completion 2017-08-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of nelfinavir | Approximately 1 year to establish MTD
  If 0/3 patients experience dose limiting toxicity, 3 patients will be treated at the next dose level. If dose limiting toxicity attributable to the study drug(s) is experienced in exactly 1/3 patients, 3 more patients (for a total of 6) will be treated at that dose level. If no additional dose limiting toxicity is observed at the expanded dose level (i.e. 1/6 with dose limiting toxicity), the dose will be escalated. Escalation will terminate as soon as two or more patients experience any dose limiting toxicity attributable to the study drug(s), at a given dose level. If 2 or more dose limiting toxicities are observed in any cohort, no further escalation will take place, and the Maximum Tolerated Dose will have been exceeded.
The toxicity of MLN9708 when combined with nelfinavir based on CTCAE grading criteria v. 4.0 | Approximately 18-24 months to observe toxicity
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI Revised Common Toxicity Criteria and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.

SECONDARY OUTCOMES:
Pharmacokinetics of both MLN9708 and nelfinavir based on parameters estimated using WinNonLin | The study as a whole is estimated to be completed in 18-24 months.
  MLN2238 concentrations-time data will be plotted on a semi-logarithmic plot and the decay of the drug concentrations over time inspected. The data will initially be analyzed using a non-compartmental and the primary pharmacokinetic parameters estimated using WinNonLin.
Pharmacodynamics of MLN9708 based on peripheral blood mononuclear cells (PBMCs) | The study as a whole is estimated to be completed in 18-24 months.
  To explore the effect of nelfinavir on the pharmacodynamics of MLN9708 (as assessed by β1 and β5 inhibition in peripheral blood mononuclear cells (PBMCs), ATF-3, CHOP and GADD34 up-regulation in PBMCs.
Pharmacodynamics of MLN9708 based on tumor tissue | The study as a whole is estimated to be completed in 18-24 months.
  To explore the effect of nelfinavir on the pharmacodynamics of MLN9708 based on tumor tissue apoptosis induction as detected by TUNEL stain, and activated caspase-3 cleavage in primary tumors.
The anti-tumor activity of the MLN9708/Nelfinavir | The study as a whole is estimated to be completed in 18-24 months.
  Disease assessments, including radiological imagining will occur initially after 9 weeks of therapy and then every 6 weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel D Lewis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States